CLINICAL TRIAL: NCT04253236
Title: A Phase 2, Multicenter, Non-Randomized, Open-Label Study of RVT-1401 for the Treatment of Patients With Warm Autoimmune Hemolytic Anemia
Brief Title: To Assess the Efficacy and Safety of RVT-1401 in the Treatment of Warm Autoimmune Hemolytic Anemia (ASCEND-WAIHA).
Acronym: ASCEND-WAIHA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RVT-1401-2003
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Results first posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Warm Autoimmune Hemolytic Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Dosing Regimen A - 680 mg weekly for 12 weeks via once weekly subcutaneous (SC) injections
  Interventions: Drug: RVT-1401 680 mg/weekly
- Cohort 2 (Experimental): Dosing Regimen B - 340 mg weekly for 12 weeks via once weekly subcutaneous (SC) injections
  Interventions: Drug: RVT-1401 340 mg/weekly

INTERVENTIONS:
Drug: RVT-1401 680 mg/weekly — Non-randomized subjects will receive subcutaneous injection of 680 mg weekly for 12 weeks of RVT-1401
  Arms: Cohort 1
Drug: RVT-1401 340 mg/weekly — Non-randomized subjects will receive subcutaneous injection of 340 mg weekly for 12 weeks of RVT-1401
  Arms: Cohort 2

SUMMARY:
This is a Phase 2 non-randomized, open-label study to investigate the efficacy, safety and tolerability of RVT-1401 in patients with Warm Autoimmune Hemolytic Anemia.

DETAILED DESCRIPTION:
This is a Phase 2, non-randomized, sequential, open-label study to investigate the safety, tolerability, PK, PD, and efficacy of RVT-1401 (680 mg/weekly and 340 mg/weekly) in patients with Warm Autoimmune Hemolytic Anemia that is worsening or refractory in spite of therapy with steroids and or immunosuppressants or worsening with steroid or immunosuppressant taper. Two cohorts of participants will be enrolled in a non-randomized sequential approach. Participants will be enrolled into Cohort 1 (680 mg/weekly) first followed by Cohort 2 (340 mg/weekly).

Following the initial dose at the Baseline Visit (Week 1, Day 1), study visits will occur weekly throughout the treatment period. Following the final dose at Week 12, visits will occur weekly through Week 14 and then at Week 16 and Week 20. Safety, PK, PD, and clinical assessments will be collected throughout the study.

Each participant will participate in the study for up to approximately 24 weeks: up to a 4-week screening period, a 12-week treatment period, and an 8-week follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Diagnosis of primary or secondary WAIHA as documented by a positive direct antiglobulin test (DAT) specific for anti-IgG alone or anti-IgG plus C3d.
3. Secondary WAIHA may only include Stage 0 chronic lymphocytic leukemia (CLL) in which separate treatment is not indicated, nor anticipated to require active management for the duration of the study.
4. Have failed or not tolerated at least one prior WAIHA treatment regimen as per local standards (e.g., steroids, rituximab, azathioprine, cyclophosphamide, cyclosporine, mycophenolate mofetil (MMF), danazol, or vincristine). Failure is defined as worsening or refractory disease despite steroids and or immunosuppressants.
5. Participants with splenectomy ≥3 months from Day 1 who are up to date on vaccinations (based on age and local guidance) are allowed.
6. At Screening and Baseline, subject's hemoglobin level must be <10 g/dL and the subject must have documented symptoms related to anemia (e.g., weakness, dizziness, fatigue, shortness of breath, chest pain).
7. Subject's concurrent treatment for WAIHA may consist only of steroids (stable dose for at least two weeks prior to Day 1), immunosuppressant therapy (azathioprine, MMF, or cyclosporine) that has been at a stable dose for at least four weeks prior to Day 1, or erythropoietin (stable dose for at least 6 weeks prior to Day 1). [Note: starting doses of WAIHA therapy must be maintained throughout the study except in the case of a rescue medication as per local standards for safety. Steroid taper down to 10 mg/day will be allowed for participants who achieve response for at least 2 weeks.]
8. A female participant is eligible to participate if she is of:

   1. Non-childbearing potential defined as pre-menopausal females with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy; hysteroscopic sterilization, or postmenopausal defined as 12 months of spontaneous amenorrhea.
   2. Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or Principal Investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female participants must agree to use contraception until 90 days after the last dose of study treatment.
9. Male participants must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study treatment until 90 days after the last dose of study treatment.
10. Willing and capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Other, more specific inclusion criteria are defined in the protocol.

Exclusion Criteria:

1. Participants with other types of AIHA (e.g., cold antibody AIHA, cold agglutinin syndrome, mixed type AIHA, or paroxysmal cold hemoglobinuria).
2. Participants requiring more than 2 units of RBC per week in the 2 weeks prior to Screening and Baseline.
3. Use of rituximab, any monoclonal antibody for immunomodulation, or proteasome inhibitor, within the past 3 months prior to Screening.
4. Immunoglobulins given by SC, IV (IVIG), or intramuscular route, or plasmapheresis/plasma exchange (PE) within 60 days before Screening.
5. Total IgG level <6 g/L (at Screening).
6. Absolute neutrophil count <1000 cells/mm3(at Screening).

Other, more specific exclusion criteria are defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (5):
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital Cancer Center - Hematology/Oncology, Boston, Massachusetts
  - University of Michigan - Internal Medicine Division of Hematology/Oncology, Ann Arbor, Michigan
  - Leo W. Jenkins Cancer Center, Greenville, North Carolina
- Israel (3):
  - Ha'Emek Medical Center, Afula
  - Carmal MC, Haifa
  - Meir Medical Center, Kfar Saba
- South Korea (6):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital - Department of Internal Medicine, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hospital Universitario Quirónsalud Madrid, Barcelona
  - Hospital Universitario Quirón, Madrid
- Thailand (4):
  - Faculty of Medicine, Chulalongkorn University, King Chulalongkorn Memorial Hospital, Bangkok
  - Faculty of Medicine, Chiang Mai University, Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Faculty of Medicine, Prince of Songkla University,Songklanagarind Hospital, Hat Yai
  - Faculty of Medicine, Khon Kaen University, Srinagarind Hospital, Khon Kaen
- Royal Cornwall Hospital, Truro, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 11 participants were screened, of which 5 participants were enrolled and randomized into the study. The study was terminated early prior to completion of dosing all participants in Cohort 1 and prior to initiating Cohort 2, as efficacy and safety conclusions could not be drawn and Pharmacokinetics/Pharmacodynamics (PK/PD) data were limited, due to the small number of participants (n=5) enrolled in the study.
Groups:
- Cohort 1: RVT-1401 680 mg/Week: Participants received RVT-1401 680 milligram (mg) subcutaneous (SC) injection weekly for 12 weeks.
- Cohort 2: RVT-1401 340 mg/Week: Participants were planned to receive RVT-1401 340 mg SC injection weekly for 12 weeks.
Period: Overall Study
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Started | 5 | 0
Completed | 2 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Safety Concerns | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least one dose of study treatment. Only data for Cohort 1 is presented as study was terminated early prior to completion of dosing all participants in Cohort 1 and and Cohort 2 was not initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders at Week 13
Description: Responders were defined as the participants with level of hemoglobin (Hb) >=10 grams per deciliter (g/dL) with at least a >=2 g/dL increase from Baseline without rescue therapy or blood transfusions in the previous two weeks.
Time Frame: Week 13
Population: Safety population: All participants who enrolled in the study and received at least 1 dose of study treatment. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Participants | 1 |

2. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Serious AE (SAE), Treatment-related Adverse Event (AE), and Death
Description: AEs were defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Clinically significant changes determined by the Investigator such as vital signs, Electrocardiograms (ECGs), and clinical laboratory values were also reported as AEs. TEAEs were defined as AEs that either started on or after the date of the first dose of study drug. SAEs were defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event that may have jeopardized the participant or may have required medical or surgical intervention to prevent one of the other outcomes listed in the definition.
Time Frame: Up to Week 20
Population: Safety Population. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Participants
  TEAEs | 5 |
  SAEs | 1 |
  Treatment-related AEs | 4 |
  Deaths | 0 |

3. Secondary Outcome: Time to Response
Description: The time to response was defined as the amount of time to achieve response (Hb levels >=10 g/dL with at least a >=2 g/dL increase from Baseline without rescue therapy or blood transfusions in the previous 2 weeks).
Time Frame: Up to Week 13
Population: Safety Population. Only those participants with data available at the specified time points were analyzed. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Number; unit: Weeks
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 1 | 0
Weeks | 3 |

4. Secondary Outcome: Time to Achieving Hb Levels in the Normal Range
Description: Time to achieving Hb levels in the normal range was assessed.
Time Frame: Up to Week 13
Population: as for outcome 3
Measure: Number; unit: Weeks
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 1 | 0
Weeks | 5 |

5. Secondary Outcome: Number of Participants With Change in Functional Assessment of Chronic Illness Therapy-fatigue (FACIT-F) Score
Description: The FACIT-F scale was a validated scale which measured the physical, emotional and social implications of fatigue, one of the key clinical manifestations of warm autoimmune hemolytic anemia. Scores ranged from 0-52, a higher score indicated a higher quality of life. A score of less than 30 indicated severe fatigue. The scale took approximately 5-10 minutes to complete.
Time Frame: Up to Week 13
Population: Safety Population. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Participants | 3 |

6. Secondary Outcome: Number of Participants With Change in Medical Research Council (MRC) Breathlessness Scale
Description: The MRC Breathlessness scale is a questionnaire that consisted of 5 statements about perceived Breathlessness and the focus of the scale was to quantify the disability associated with breathlessness. Score ranged from Grade 0 (limited to no disability) to Grade 4 (severe disability); higher score indicated severe disability.
Time Frame: Up to Week 13
Population: Safety Population. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Participants | 4 |

7. Secondary Outcome: Number of Participants With Change in Euro Quality-5 Dimension-3 Level (EQ-5D-3L) Score
Description: The EQ-5D-3L is a validated measurement of health-related quality of life. The scale consists of 2 components, the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The descriptive system evaluates mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1=no problems, 2=some problems, and 3=extreme problems; a lower score indicated better quality of life. The EQ VAS records the participant's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' (100) and 'Worst imaginable health state' (0).
Time Frame: Up to Week 20
Population: Safety Population. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Participants | 4 |

8. Secondary Outcome: Concentration of RVT-1401 Pre-dose
Description: Blood samples were planned to be collected at indicated time points to measure the concentration of RVT-1401 pre-dose (Ctrough) as an assessment of the pharmacokinetic (PK) RVT-1401.
Time Frame: Pre-dose, Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12 and 13 post-dose
Population: Safety Population. Data could not be calculated for Cohort 1 due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed). Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams per liter
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Milligrams per liter | NA (NA) — Data could not be calculated due to high proportion of non-quantifiable values (>30% of values were imputed). |

9. Secondary Outcome: Number of Participants With Presence of Anti-RVT 1401 Antibodies
Description: Blood samples were collected at indicated time points to determine presence of anti-RVT 1401 antibodies. Participants with presence of anti-RVT 1401 antibodies is reported
Time Frame: Pre-dose on Weeks 1, 3, 5, 8, 13 and Week 20
Population: Safety population. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Participants | 0 |

10. Secondary Outcome: Number of Participants With Change in Levels of Total Immunoglobulin (Ig)G and IgG Subclasses (1-4)
Description: Blood samples were collected at indicated time points for pharmacodynamic (PD) analysis of serum total IgG and IgG subclasses (1-4) concentrations. Participants with changes in levels of Total IgG and IgG Subclasses (1-4) is reported.
Time Frame: Up to Week 20
Population: Safety Population. Data was not collected for Cohort 2 due to early termination of the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
Number analyzed (Participants) | 5 | 0
Participants
  Total IgG | 5 |
  IgG Subclasses (1-4) | 5 |

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious TEAEs and SAEs were collected up to Week 20 in Cohort 1.
Description: Safety Population. Only data for Cohort 1 is presented as the study was terminated in Part 1; hence, Cohort 2 was not initiated.
Arm/Group | Cohort 1: RVT-1401 680 mg/Week | Cohort 2: RVT-1401 340 mg/Week
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 5/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: RVT-1401 680 mg/Week (N=5) | Cohort 2: RVT-1401 340 mg/Week (N=0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: RVT-1401 680 mg/Week (N=5) | Cohort 2: RVT-1401 340 mg/Week (N=0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT04253236/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT04253236/SAP_001.pdf